CLINICAL TRIAL: NCT07140523
Title: A Multicenter, Randomized, Open-Label, Blinded Endpoint Evaluation, Active Controlled Study to Compare the Efficacy and Safety of SRSD107 and Enoxaparin in Adult Subjects Undergoing Elective Primary Unilateral Total Knee Arthroplasty
Brief Title: A Study to Compare the Efficacy and Safety of SRSD107 and Enoxaparin in Adult Subjects Undergoing TKA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sirius Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SRSD107-201
Record Dates: First submitted 2025-08-11; First posted 2025-08-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SRSD107 low dose (Experimental): Cohort 1: SRSD107, low dose level, subcutaneous (s.c.), single dose
  Interventions: Drug: SRSD107
- SRSD107 medium dose (Experimental): Cohort 2: SRSD107, medium dose level, subcutaneous (s.c.), single dose
  Interventions: Drug: SRSD107
- SRSD107 high dose (Experimental): Cohort 3: SRSD107, high dose level, subcutaneous (s.c.), single dose
  Interventions: Drug: SRSD107
- Enoxaparin (Active Comparator): Cohort 4: Enoxaparin 40 mg s.c., once a day (q.d.), 12 ±2 days post-surgery
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: SRSD107 — SRSD107 is an investigational siRNA product for anticoagulants.
  Arms: SRSD107 high dose; SRSD107 low dose; SRSD107 medium dose
Drug: enoxaparin — Enoxaparin is a low molecular weight heparin [LMWH] indicated for Prophylaxis of deep vein thrombosis (DVT) in abdominal surgery, hip replacement surgery, knee replacement surgery, or medical patients with severely restricted mobility during acute illness.
  Other Names: Clexane; Lovenox
  Arms: Enoxaparin

SUMMARY:
This is a Phase 2, multicenter, randomized, open-label, parallel group, blinded endpoint evaluation, active-controlled, dose-finding study.This study is designed to compare the efficacy and safety of 3 dose levels of SRSD107 and enoxaparin 40 mg daily in subjects undergoing elective primary unilateral TKA.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy and safety of 3 dose levels of SRSD107 and enoxaparin 40 mg daily in subjects undergoing elective primary unilateral TKA. While the identity of the study drug will be unblinded, the specific dose of SRSD107 will be blinded. Up to approximately 450 subjects will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent before any study assessment is performed.
2. Male and female subjects, of any race, between 60 and 80 years of age, inclusive.
3. Body mass index between 18.0 and 35.0 kg/m2, inclusive.
4. Eligible to undergo elective primary unilateral TKA under general anesthesia.
5. Willing to comply with study requirements including taking study drug at least 28 days prior to TKA, clinic visits, and venography at 10-14 days post TKA.
6. aPTT, PT, and INR within the normal reference range at screening.

Exclusion Criteria:

1. Active bleeding requiring medical or surgical intervention within 4 weeks prior to screening.
2. Known bleeding disorder; history of increased bleeding tendency or any other condition that in the opinion of the investigator contraindicates prophylactic anticoagulation.
3. History of intracranial, intraspinal, or intraocular bleeding.
4. Evidence of active cancer, or a history of malignancy, within 2 years prior to screening.
5. Myocardial infarction, DVT, PE, stroke , transient ischemic attack, systemic embolism, valvular thrombosis, or splanchnic thrombosis in the 6 months prior to screening.
6. Uncontrolled blood pressure at the time of screening.
7. Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2.
8. Liver dysfunction, liver cirrhosis, history of hepatic encephalopathy, esophageal varices, or portocaval shunt.
9. Clinically significant anemia at screening.
10. Platelet counts <100,000/m3 at screening or a history of heparin-induced thrombocytopenia.
11. Positive test for human immunodeficiency virus (HIV) , positive hepatitis B surface antigen, and/or active hepatitis C at screening.
12. Ongoing or anticipated need for anticoagulation or antiplatelet therapy from 7 days prior to surgery through the EoS visit.
13. Participation in an interventional clinical study within 5 half-lives of the investigational drug or 30 days prior to screening, whichever is longer.
14. Use of any ASO or siRNA products within 1 year prior to screening. Diet and Lifestyle.
15. Recent or current history of alcoholism or recreational drug abuse.
16. History of hypersensitivity to any of the study drugs or its excipients, to drugs of similar chemical classes or drugs issued from the same biologic origin or any contraindication listed in the label for enoxaparin.
17. Unable to undergo venography due to a known allergy to the contrast agent, anticipated poor venous access, impaired renal function, or any other reason identified and specified by the investigator.
18. Anticipated elective surgery during the study period.
19. Any other condition or circumstance that would affect the subject's ability to be compliant with study drug administration or study procedures, in the opinion of the investigator.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of total venous thromboembolism (VTE) events | From the date of surgery through 12±2 days after surgery.
  Defined as deep vein thrombosis (DVT) (asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic), non-fatal and fatal PE, and unexplained death for which PE cannot be excluded.

SECONDARY OUTCOMES:
Incidence of major VTE | From the date of surgery through 12±2 days after surgery and Day 64, respectively.
  Defined as objectively confirmed symptomatic DVT and PE, asymptomatic proximal DVT (confirmed by venogram), fatal PE, and unexplained death for which PE cannot be excluded.
Incidence of total VTE events | From the date of surgery through Day 64.
  Defined as symptomatic DVT, asymptomatic DVT (confirmed by venogram), non-fatal and fatal PE, unexplained death for which PE cannot be excluded.
Incidence of total VTE events for each individual dosing cohort of SRSD107 compared to enoxaparin | From the date of surgery through 12±2 days after surgery.
  Defined as symptomatic DVT, asymptomatic DVT (confirmed by venogram), non-fatal and fatal PE, unexplained death for which PE cannot be excluded.
Incidence of composite of major bleeding (MB) and clinically relevant non-major bleeding (CRNMB) | From the Pre-surgical Period through 12±2 days after surgery.
  Based on the 2013 Guideline on clinical investigation of medicinal products for prevention of venous thromboembolism (VTE) in patients undergoing high VTE-risk surgery (EMA/CHMP/325170/2012), as well as updated guidance from the International Society of Thrombosis and Haemostasis (ISTH; Schulman 2010).
Incidence of composite of MB, CRNMB, and any bleeding | From the Pre-surgical Period through 12±2 days after surgery, Day 64, and Day 169, respectively.
  Based on the 2013 Guideline on clinical investigation of medicinal products for prevention of venous thromboembolism (VTE) in patients undergoing high VTE-risk surgery (EMA/CHMP/325170/2012), as well as updated guidance from the International Society of Thrombosis and Haemostasis (ISTH; Schulman 2010).
Incidence of MB | From the Pre-surgical Period through 12±2 days after surgery.
  Based on the 2013 Guideline on clinical investigation of medicinal products for prevention of venous thromboembolism (VTE) in patients undergoing high VTE-risk surgery (EMA/CHMP/325170/2012), as well as updated guidance from the International Society of Thrombosis and Haemostasis (ISTH; Schulman 2010).
Incidence of CRNMB | From the Pre-surgical Period through 12±2 days after surgery.
  Based on the 2013 Guideline on clinical investigation of medicinal products for prevention of venous thromboembolism (VTE) in patients undergoing high VTE-risk surgery (EMA/CHMP/325170/2012), as well as updated guidance from the International Society of Thrombosis and Haemostasis (ISTH; Schulman 2010).
Incidence of adverse events (AEs) | From Day 1 through Day 169.
  An adverse event (AE) is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nové Město na Moravě, Nové Město na Moravě, Czechia

IPD SHARING:
Plan to Share IPD: No